CLINICAL TRIAL: NCT02046135
Title: Sodium Bicarbonate to Prevent Acute Kidney Injury in Children Undergoing Cardiac Surgery: A Randomized Clinical Trial
Brief Title: Sodium Bicarbonate to Prevent Acute Kidney Injury in Children Undergoing Cardiac Surgery
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Statistical analysis at interim analysis determined futility in continuing.
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, James Schneider, Fellowship Director Critical Care, Northwell Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 13-007B
Record Dates: First submitted 2014-01-22; First posted 2014-01-27 (Estimated); Results first posted 2020-12-28 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Acute Kidney Injury; Congenital Heart Disease
Keywords: Pediatric; Sodium bicarbonate; Acute kidney injury; Cardiac surgery
MeSH Terms: conditions — Acute Kidney Injury; Heart Defects, Congenital | interventions — Sodium Bicarbonate; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sodium bicarbonate (Experimental): At the start of the surgery, the patient will receive NaHCO3 as a continuous infusion of D5% 1/3NS + 100 meq/L NaHCO3 + 20 meq/L KCl at maintenance IVF (solution contains ~154 meq of sodium which is equivalent to normal saline). The NaHCO3 infusion will continue for the first 24 hours after the discontinuation of CPB. After 24 hours of receiving the NaHCO3 infusion, the IVF administered to the patient will be the standard solutions used in the PICU at CCMC.
  Interventions: Drug: Sodium Bicarbonate
- Sodium Chloride (Active Comparator): At the start of surgery, patients in the control arm will receive D5% Normal Saline + 20 meq/L KCl at maintenance IVF. After 24 hours, standard IVF, not containing NaHCO3 or Na acetate will be administered for the duration of the PICU stay as required, determined by the clinicians primarily caring for the patient postoperatively.
  Interventions: Drug: Sodium Chloride

INTERVENTIONS:
Drug: Sodium Bicarbonate
  Arms: Sodium bicarbonate
Drug: Sodium Chloride
  Arms: Sodium Chloride

SUMMARY:
The proposed study will investigate the effect of sodium bicarbonate on the prevention of acute kidney injury in children undergoing cardiac surgery with cardio-pulmonary bypass. The investigators hypothesize that the occurrence of acute kidney injury will be less in children treated with sodium bicarbonate in the perioperative period when compared to placebo. The specific aims of this proposal are as follows:

1. To institute a prospective, randomized, double-blinded, placebo-controlled trial in pediatric subjects undergoing cardiac surgery to determine the efficacy of sodium bicarbonate on prevention of acute kidney injury as measured by pRIFLE criteria. 2. To examine whether treatment with sodium bicarbonate modifies the duration of acute kidney injury, fluid balance, hospital length of stay, need for dialysis, and progression to kidney failure. 3. To determine the relevance of NGAL as a biomarker to predict development of acute kidney injury.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects age ≤18 years
2. Subjects scheduled for cardiac surgery with cardiopulmonary bypass

Exclusion Criteria:

1. Subjects with abnormal creatinine clearance (<90 ml/min/1.7m2) as measured by the Schwartz formula
2. Subjects with known cystic kidney disease or posterior ureteral valves (subjects with solitary kidney, single multicystic/dysplastic kidney, hydronephrosis will not be excluded if renal function is preserved)
3. Subjects with known metabolic disorder
4. Premature infants born <30 weeks gestation and <30 days old due to risk of intraventricular hemorrhage

Subjects in severe cardiogenic shock post-operative requiring extra-corporeal membrane oxygenation (ECMO) or left ventricular assist device (LVAD) will be withdrawn from the study.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 51 (Actual)
Dates: Start 2013-09; Primary Completion 2017-06 (Actual); Study Completion 2017-07-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Schneider, MD, Principal Investigator — Cohen Children's Medical Center of New York
Locations (1):
- Cohen Children's Medical Center of New York, New Hyde Park, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Sodium Bicarbonate: At the start of the surgery, the patient will receive NaHCO3 as a continuous infusion of D5% 1/3NS + 100 meq/L NaHCO3 + 20 meq/L KCl at maintenance IVF (solution contains ~154 meq of sodium which is equivalent to normal saline). The NaHCO3 infusion will continue for the first 24 hours after the discontinuation of CPB. After 24 hours of receiving the NaHCO3 infusion, the IVF administered to the patient will be the standard solutions used in the PICU at CCMC.
  Sodium Bicarbonate
- Sodium Chloride: At the start of surgery, patients in the control arm will receive D5% Normal Saline + 20 meq/L KCl at maintenance IVF. After 24 hours, standard IVF, not containing NaHCO3 or Na acetate will be administered for the duration of the PICU stay as required, determined by the clinicians primarily caring for the patient postoperatively.
  Sodium Chloride
Period: Overall Study
Arm/Group | Sodium Bicarbonate | Sodium Chloride
Started | 26 | 25
Completed | 26 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sodium Bicarbonate | Sodium Chloride | Total
Number analyzed (Participants) | 26 | 25 | 51
Age, Continuous [Median (Inter-Quartile Range); unit: months] | 4.5 [1.8 to 10.3] | 5 [2 to 52.5] | 5 [2 to 27]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 26
  Male | 13 | 12 | 25
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Height [Median (Inter-Quartile Range); unit: centimeters] | 60.5 [52 to 72.1] | 62 [51 to 107.9] | 61.6 [51.8 to 88.1]
Weight [Median (Inter-Quartile Range); unit: kg] | 6 [3.5 to 8.6] | 5.8 [3.9 to 16.1] | 5.9 [3.7 to 12.1]

OUTCOME MEASURES:

1. Primary Outcome: Acute Kidney Injury
Description: The number of patients who developed AKI in each arm of the study. AKI was measured by the Pediatric Risk, Failure, Loss of Function, and End-Stage Renal Disease (pRIFLE) criteria or an absolute increase in creatinine of 0.3mg/dl.
Time Frame: 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Sodium Bicarbonate | Sodium Chloride
Number analyzed (Participants) | 26 | 25
Participants | 19 | 20

2. Secondary Outcome: Cumulative Fluid Balance
Description: Cumulative fluid balance in milliliters- comparison of all fluid intake vs all fluid output from the time of ICU admission post-operatively for the first 6 days post-operatively or until the time of discharge, whichever came first.
Time Frame: 6 days
Measure: Median (Inter-Quartile Range); unit: mL
Arm/Group | Sodium Bicarbonate | Sodium Chloride
Number analyzed (Participants) | 26 | 25
mL | -13.8 [-219.4 to 130.8] | -12.4 [-277.8 to 69]

3. Secondary Outcome: Hospital and Intensive Care Unit Length of Stay
Description: Hospital and intensive care unit length of stay in days
Time Frame: 1 month
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Sodium Bicarbonate | Sodium Chloride
Number analyzed (Participants) | 26 | 25
days | 7.5 [4.4 to 16.1] | 7.3 [4.4 to 14.1]

4. Secondary Outcome: Need for Dialysis
Description: Need for dialysis: yes/no
Time Frame: 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | Sodium Bicarbonate | Sodium Chloride
Number analyzed (Participants) | 26 | 25
Participants | 0 | 0

5. Secondary Outcome: Length of Mechanical Ventilation
Description: Length of mechanical ventilation in days
Time Frame: 1 month
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Sodium Bicarbonate | Sodium Chloride
Number analyzed (Participants) | 26 | 25
days | 3.8 [1.2 to 6.8] | 1.2 [1.1 to 2.1]

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Sodium Bicarbonate | Sodium Chloride
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/25
Other Adverse Events (participants affected / at risk) | 0/26 | 0/25

LIMITATIONS AND CAVEATS:
Early termination leading to small number of subjects analyzed. This may lead to unreliable or uninterpretable data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2013-06-15): https://cdn.clinicaltrials.gov/large-docs/35/NCT02046135/Prot_SAP_000.pdf
  • Informed Consent Form (2013-07-15): https://cdn.clinicaltrials.gov/large-docs/35/NCT02046135/ICF_001.pdf